CLINICAL TRIAL: NCT02439125
Title: Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, 4-way Crossover, Dose-finding Study, of Eltoprazine Safety, Tolerability and Efficacy in the Treatment of Levodopa-induced Dyskinesia in Patients With Parkinson's Disease
Brief Title: A Study of Efficacy and Safety of Eltoprazine HCl for Treating Levodopa-induced Dyskinesia in Parkinson's Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amarantus BioScience Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AMBS-ELTO-201
Record Dates: First submitted 2015-04-13; First posted 2015-05-08 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease; Dyskinesia
Keywords: levodopa; dyskinesia; parkinsons disease; PD
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eltoprazine HCl 2.5 mg (Experimental): Eltoprazine HCl 2.5 mg capsules to be taken orally b.i.d. (ie, 5 mg/day) for 3 weeks
  Interventions: Drug: Eltoprazine HCl
- Eltoprazine HCl 5.0 mg (Experimental): Eltoprazine HCl 5.0 mg capsules to be taken orally b.i.d. (ie, 10 mg/day) for 3 weeks
  Interventions: Drug: Eltoprazine HCl
- Eltoprazine HCl 7.5 mg (Experimental): Eltoprazine HCl 7.5 mg capsules to be taken orally b.i.d. (ie, 15 mg/day) for 3 weeks
  Interventions: Drug: Eltoprazine HCl
- Placebo (Placebo Comparator): Placebo capsules to be taken orally b.i.d. for 3 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltoprazine HCl — 2.5 mg b.i.d. orally for 3 weeks
  Arms: Eltoprazine HCl 2.5 mg
Drug: Eltoprazine HCl — 5.0 mg b.i.d. orally for 3 weeks
  Arms: Eltoprazine HCl 5.0 mg
Drug: Eltoprazine HCl — 7.5 mg b.i.d. orally for 3 weeks
  Arms: Eltoprazine HCl 7.5 mg
Drug: Placebo — b.i.d. orally for 3 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of eltoprazine to treat levodopa-induced dyskinesia in patients with Parkinson's disease

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, crossover, dose-range finding study in patients with Parkinson's disease and levodopa-induced dyskinesia. The study will examine the effects of three different doses of eltoprazine HCl, compared to placebo, on severity of dyskinesia, parkinsonian symptoms, patient function, safety and tolerability, using Parkinson's disease rating scales, patient diaries and physiological measurement of abnormal movement by means of motion sensors.

ELIGIBILITY:
Inclusion Criteria:

* outpatient with idiopathic PD
* stable dose of anti-parkinsonian medication for at least four weeks before the Screening Visit
* daily levodopa dose ≥300 mg per day divided into at least three doses
* treated with levodopa for at least three years prior to study entry
* moderate to severely disabling levodopa-induced dyskinesia for at least three months prior to study entry
* dyskinesia for, on average, >25% of the waking day

Exclusion Criteria:

* inability to use the motion sensors or electronic diaries correctly
* surgical treatment for PD, e.g. Deep Brain Stimulation, within the last six months or planned during the study
* unstable co-existing psychiatric disease including psychosis, depression or cognitive impairment
* Mini Mental State Examination score of <24
* moderate or severe renal, or severe hepatic, impairment
* treatment with selective serotonin re-uptake inhibitors (SSRI) or any combined serotonin-norepinephrine re-uptake inhibitors (SNRI), such as tryptizol, citalopram, escitalopram, sertraline, mianserin, mirtazapin, paroxetin, venlafaxine and St John's Wort, within four weeks prior to the Screening Visit
* treatment with medications with the potential for drug-interactions (MAO-A inhibitors, apomorphine, aripiprazol, carbamazepine, clozapine, phenytoin, tramadol, quetiapine, varfaine, valproic acid). Patients taking amantadine will comprise no more than 25% of the study population
* current history of a clinically significant and uncontrolled medical condition that may affect the safety of the patient or preclude adequate participation in the study
* pregnant or breast-feeding
* received any other investigational medicinal product within 30 days of Screening

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical impact of dyskinesia measured by total UDysRS (Unified Dyskinesia Rating Scale) score | 84 days
  Clinical impact on dyskinesia measured by total UDysRS (Unified Dyskinesia Rating Scale) score at the end of each Treatment Period on Days 21, 42, 63 and 84

SECONDARY OUTCOMES:
• PD motor symptoms assessed by MDS-UPDRS, diaries and physiological measurement with motion sensor system | 84 days
  • PD motor symptoms assessed by MDS-UPDRS, diaries and physiological measurement with motion sensor system
Dyskinesia severity using physiological motion sensor system | 84 days
  Dyskinesia severity using physiological motion sensor system
Patient function using MDS-UPDRS and UDysRS questionnaires quantify dyskinesia and Parkinsonian motor symptoms. | 84 days
  Patient function using MDS-UPDRS and UDysRS questionnaires
Safety and tolerability: adverse events, physical and neurological exams, safety laboratory values, vital signs and ECG | 94 days
  Safety and tolerability: adverse events, physical and neurological exams, safety laboratory values, vital signs and ECG

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Keywood, MBBS,MRCP,, Study Director — Amarantus BioScience Holdings, Inc.
Locations (1):
- Parkinson's Disease and Movement Disorders Center, Boca Raton, Boca Raton, Florida, United States

REFERENCES:
- [Result] Svenningsson P, Rosenblad C, Af Edholm Arvidsson K, Wictorin K, Keywood C, Shankar B, Lowe DA, Bjorklund A, Widner H. Eltoprazine counteracts l-DOPA-induced dyskinesias in Parkinson's disease: a dose-finding study. Brain. 2015 Apr;138(Pt 4):963-73. doi: 10.1093/brain/awu409. Epub 2015 Feb 10. PMID 25669730
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217
- See also: Related Info — http://foxtrialfinder.michaeljfox.org/